CLINICAL TRIAL: NCT06526117
Title: Primary Prevention of Stroke in Children With SCD in Sub-Saharan Africa II: A Multicenter, Open-label, Single-arm Type I Hybrid Clinical Trial
Brief Title: Stroke Prevention in Nigeria 2 Trial
Acronym: SPRING-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Aminu Kano Teaching Hospital (Other); Murtala Muhammed Specialist Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Michael DeBaun, Professor, Vice Chair, Chair, Clinical Research, Director, Vanderbilt/Meharry Center of SCD, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 231110; U01NS129143 (NIH)
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Sickle Cell Disease; Stroke
Keywords: primary stroke prevention; hydroxyurea; low income country; sub-Saharan Africa
MeSH Terms: conditions — Anemia, Sickle Cell; Stroke | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low or Moderate Dose Hydroxyurea (Experimental): Initial treatment with Hydroxyurea at 10 mg/kg/day (range 7 to 15 mg/kg/day) for primary stroke prevention. Subsequent treatment with moderate-dose hydroxyurea (20 mg/kg/day (range 17.5 - 26 mg/kg/day)) based after at least two severe pain events requiring physician contact during the trial.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — The study intervention will include initial treatment with low-dose hydroxyurea therapy at 10 mg/kg/day (range 7 - 15 mg/kg/day), with subsequent increase to moderate dose hydroxyurea therapy at 20 mg/kg/day (range 17.5 - 26 mg/kg/day) after at least two severe events requiring physician contact.
  Other Names: Hydrea

SUMMARY:
The primary goal of this study is to complete a multicenter single-arm, type I hybrid trial to assess the effectiveness of hydroxyurea therapy for primary stroke prevention in high-risk children with sickle cell anemia (SCA) living in Nigeria in routine care settings.

DETAILED DESCRIPTION:
Strokes in sickle cell anemia (SCA), particularly in children living in Africa, are associated with significant morbidity and an increased risk of premature death. In the US, primary stroke prevention in children with SCA involves screening for elevated Transcranial Doppler ultrasound (TCD) velocity coupled with regular blood transfusion therapy for persons with elevated velocities. However, regular blood transfusion therapy is not a viable option for children with SCA in Nigeria for several reasons, including 1) inadequate supply of blood (still donor exchange system; 2) availability and cost of monthly blood transfusions for preventive therapy as opposed to emergency therapy; 3) unsafe blood supplies with a high probability of blood-borne infections and alloimmunization; and 4) children that receive regular blood transfusion will ultimately require daily iron chelation an unaffordable undertaking in low-income countries.

This multicenter open-label, single-arm type I hybrid trial will assess the effectiveness of Hydroxyurea therapy for primary stroke prevention in children with sickle cell anemia (SCA) living in Nigeria. A recently completed double-blind, parallel-group phase III randomized controlled trial (SPRING), involved comparing low-dose to moderate-dose hydroxyurea for primary stroke prevention in children with SCA and abnormal transcranial Doppler (TCD) velocities (>200 cm/sec). Children with abnormal TCD velocities have a high stroke risk of approximately 10.7 events per 100 person-years (observation arm in the STOP trial). In the low- (n=109) and moderate-dose (n=111) hydroxyurea groups, the stroke incidence rates were 1.2 and 1.9 per 100 person-years, respectively, p=0.77 (combined incidence rate 1.5 per 100 person-years). Despite equal efficacy for stroke prevention in both treatment groups, moderate- when compared to low-dose hydroxyurea, was more effective in preventing severe acute pain and all-cause hospitalizations. Our findings supported the American Society of Hematology's evidence-based guidelines for hydroxyurea therapy for primary stroke prevention in low-income settings. The hypothesis to be tested in the SPRING-2 study is in a multicenter single-arm type I hybrid trial, for children with abnormal TCD velocities treated with hydroxyurea, the stroke incidence rate will be non-inferior to the SPRING trial results, with an upper non-inferiority margin of 4 strokes per 100-person-years. The point estimate method was used to determine the non-inferiority margin based on the Nigerian pediatrician's judgment of what maximum stroke rate would be clinically meaningful to demonstrate the effectiveness and justify treatment for the high-risk stroke group. A non-inferiority test with an overall sample size of 220 will achieve 91% power at a 0.050 significance level to detect non-inferiority when the expected proportion of strokes is 0.035, a minimum follow-up period of 2.5 years and a loss to follow-up of 10% per year. The study will follow standard of care procedures, including clinic visits every 3 months and complete blood cell counts every 6 months. The following aims will be conducted as part of the trial: 1) Determine the incidence of the first stroke in children with abnormal TCD velocities treated with hydroxyurea for 2.5 years in the type 1 hybrid trial; 2) Evaluate the implementation and sustainability of the intervention within the extended RE-AIM framework; 3) Evaluate the cost-effectiveness of low- compared to a higher dose of hydroxyurea for primary stroke prevention in children with abnormal TCD velocities. Capacity building for three Nigerian Multiple Principal Investigators, statisticians, and nurses will be focused on three areas-: 1) developing a Nigerian data coordinating center and the required skills to support a clinical trial; 2) developing a regional TCD course for nurses, enhancing task shifting and reach, and 3) performing cost-effective analysis for the type I hybrid trial comparing low-and moderate dose hydroxyurea.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the SPRING-2 Trial will consist of:

* Diagnosis of HbSS or HbSB0 confirmed by high-performance liquid chromatography (HPLC);
* Informed consent from the parent/legal guardian and assent from the patient at least 7 years of age;
* Two TCD flow velocity readings of >or equal to180 cm/sec and < 220 cm/sec or one TCD velocity reading > or equal to 220 cm/sec; typically the repeat TCD is performed on the same day so treatment can start immediately;
* Age between 5 and 12 years (assessment can take place up until the 13th birthday), which includes the peak age of onset of strokes in SCA, ~ 6 yo; and
* Ability to swallow the hydroxyurea capsule.

Exclusion Criteria:

The exclusion criteria will be the following:

* Prior stroke or TIA by history, or concern for moderate or severe neurological deficit based on a positive validated "10 questions" screening;
* Other significant organ system dysfunction or other contraindication to hydroxyurea;
* Children who are already on therapy with either blood transfusion or hydroxyurea therapy;
* Significant cytopenias (absolute neutrophil count (ANC) <1500, platelets <150,000/ul, reticulocytes <80,000/ul, unless Hb is > 9 g/dl], renal insufficiency (creatinine > 0.8 mg/dl); and
* History of seizures or diagnosis of epilepsy, and 6) metal in the body that would make MRI unsafe. The rationale for excluding children under 5 years old: Despite being a vulnerable age group for strokes, children younger than 5 years were excluded because a significant proportion of this population is unable to swallow a capsule, the only stable form of hydroxyurea available in Nigeria.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate of Clinical Stroke or TIA | 5 years
  The incidence rate of clinical stroke or TIA in participants treated with low- or moderate-dose hydroxyurea.

SECONDARY OUTCOMES:
Incidence of All-Cause Hospitalizations | 5 years
  To evaluate all-cause hospitalizations with low-dose or moderate-dose hydroxyurea during clinic visits. Participants will be interviewed to determine the number of interim hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R DeBaun, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- Nigeria (2):
  - Aminu Kano Teaching Hospital, Kano
  - Murtala Muhammad Specialist Hospital, Kano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams RJ, McKie VC, Hsu L, Files B, Vichinsky E, Pegelow C, Abboud M, Gallagher D, Kutlar A, Nichols FT, Bonds DR, Brambilla D. Prevention of a first stroke by transfusions in children with sickle cell anemia and abnormal results on transcranial Doppler ultrasonography. N Engl J Med. 1998 Jul 2;339(1):5-11. doi: 10.1056/NEJM199807023390102. PMID 9647873
- [Background] Abdullahi SU, Jibir BW, Bello-Manga H, Gambo S, Inuwa H, Tijjani AG, Idris N, Galadanci A, Hikima MS, Galadanci N, Borodo A, Tabari AM, Haliru L, Suleiman A, Ibrahim J, Greene BC, Ghafuri DL, Rodeghier M, Slaughter JC, Kirkham FJ, Neville K, Kassim A, Trevathan E, Jordan LC, Aliyu MH, DeBaun MR. Hydroxyurea for primary stroke prevention in children with sickle cell anaemia in Nigeria (SPRING): a double-blind, multicentre, randomised, phase 3 trial. Lancet Haematol. 2022 Jan;9(1):e26-e37. doi: 10.1016/S2352-3026(21)00368-9. PMID 34971579